CLINICAL TRIAL: NCT07196475
Title: Safety And Efficacy Of Transurethral Focal Laser Ablation of Prostatic Adenoma In Comparison With Transurethral Prostatectomy For Management Of Benign Prostatic Adenoma Comparative Randomized Prospective Study
Brief Title: Transurethral Focal Laser Ablation Versus Transurethral Prostatectomy For Management Of Benign Prostatic Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MD 19/2022
Record Dates: First submitted 2025-08-21; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-08

CONDITIONS: Benign Prostate Hypertrophy(BPH)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Procedure: FOCAL LASER ABLATION OF PROSTATE — All monopolar TURP procedures were performed under spinal anaesthesia, whereas all TU-FLAP procedures were conducted under local anaesthesia with intravenous sedation. A single experienced surgical team performed all operations, with each surgeon having completed over 100 similar procedures prior to the study's initiation. Prophylactic antibiotic coverage with a third-generation cephalosporin has been administered at the time of anaesthesia induction. Cases were placed in the lithotomy position, followed by diagnostic urethrocystoscopy. In the TU-FLAP group, a 980 nm diode laser fig(1) by applying end-firing fiber fig(2) was introduced via the side working channel of a 22 Fr cystoscope under local anesthesia. Laser energy was applied at 15 watts for two minutes at multiple sites within the right and left prostatic lobes, approximately 1.5 cm distal to the bladder neck, with 1 cm spacing between punctures. In cases with an enlarged median lobe, one or two additional laser punctures were

SUMMARY:
Introduction and objectives: Laser prostatectomy has become an increasingly popular and effective alternative to transurethral resection of the prostate (TURP) for the treatment of benign prostatic hyperplasia (BPH).-. This study focuses on assessing the safety, efficacy, and postoperative complications of Transurethral Focal Laser Ablation of Prostatic Adenoma (TU-FLAP) versus M-TURP in managing BPH, with a 12-month monitoring.

Patients and Methods: 60 BPH cases meeting the inclusion criteria have randomly been assigned into 2 equal groups to undergo either TU-FLAP or M-TURP. Outcomes have been assessed using IPSS, QoL, Qmax, operative time, catheterization ,duration of hospital stay, PVR, PSA, and residual prostate volume. Safety was evaluated based on perioperative and postoperative complications.

DETAILED DESCRIPTION:
INTRODUCTION Benign prostatic hyperplasia is a frequent condition between aging men, often leading to lower urinary tract symptoms (LUTS) that significantly impair quality of life. TURP was long considered the gold standard surgical intervention for prostates ranging from 30 to 80 grams [1]. Despite its efficacy, TURP is associated with notable risks, including intraoperative bleeding and the potential for fluid absorption leading to dilutional hyponatremia, commonly referred to as TUR syndrome. These risks are particularly pronounced in patients with larger prostates or those on anticoagulant therapy. Additionally, TURP requires considerable surgical expertise and is associated with a steep learning curve [2].

Transperineal focal laser ablation (TPLA) has emerged as a novel approach, targeting obstructive transitional zone tissue while sparing adjacent structures. This technique achieves debulking by inducing strategic coagulative necrosis, which is subsequently reabsorbed by the body, resulting in reduced prostate volume with minimal impact on urinary continence and sexual function [3]. Similarly, Rezūm therapy utilizes convective water vapor energy to ablate prostatic tissue. It is an office-based procedure that requires no general anesthesia and has demonstrated durable improvement in LUTS while preserving sexual function [4]. Despite these advancements, both TPLA and Rezūm are constrained by limited availability and relatively narrow indications. In this context, TU-FLAP represents a new approach. Unlike existing laser therapies, TU-FLAP is designed to ablate obstructive prostatic adenoma via a transurethral route, without disturbing the urethral mucosa or the ejaculatory ducts. This distinction provides a significant advantage in preserving antegrade ejaculation and reducing the risk of urethral trauma-outcomes often compromised in TURP, HoLEP (Holmium laser Enucleation of the prostate), and other enucleative procedures.

To the best of our knowledge, this is the 1st research to evaluate TU-FLAP using diode laser energy under local anesthesia. The technique leverages real-time endoscopic visualization to deliver precise, targeted energy into the prostatic adenoma, while avoiding direct contact with critical structures such as the urethral sphincter.

This randomized controlled trial was designed to compare TU-FLAP with monopolar TURP in terms of operative metrics, postoperative complications, and patient-reported symptom scores over a one year follow-up duration.

Preoperative workup All cases had a standardized preoperative evaluation, including the International Prostate Symptom Score (IPSS), International Index of Erectile Function (IIEF), and quality of life (QoL) assessment. Physical examination included a digital rectal examination (DRE). Additional assessments included uroflowmetry, urinalysis, and urine culture when indicated, as well as measurement of serum prostate-specific antigen (PSA). Pelvic ultrasound was performed to determine post-void residual urine (PVR), and transrectal ultrasound (TRUS) was used to estimate prostate volume.

Technique:

All monopolar TURP procedures were performed under spinal anaesthesia, whereas all TU-FLAP procedures were conducted under local anaesthesia with intravenous sedation. A single experienced surgical team performed all operations, with each surgeon having completed over 100 similar procedures prior to the study's initiation. Prophylactic antibiotic coverage with a third-generation cephalosporin has been administered at the time of anaesthesia induction. Cases were placed in the lithotomy position, followed by diagnostic urethrocystoscopy. In the TU-FLAP group, a 980 nm diode laser fig(1) by applying end-firing fiber fig (2) was introduced via the side working channel of a 22 Fr cystoscope under local anesthesia. Laser energy was applied at 15 watts for two minutes at multiple sites within the right and left prostatic lobes, approximately 1.5 cm distal to the bladder neck, with 1 cm spacing between punctures. In cases with an enlarged median lobe, one or two additional laser punctures were applied. Postoperative urethral catheterization has been maintained for three to seven days, depending on the volume of treated prostatic tissue and the period of preoperative urinary retention.

Postoperative Follow-up Protocol:

Efficacy was evaluated using the following parameters: International Prostate Symptom Score (IPSS), quality of life (QoL) score, operative time, maximum urinary flow rate (Qmax), , length of hospital stay, duration of catheterization, post-void residual urine volume (PVR), serum prostate-specific antigen (PSA), and residual prostate volume measured via transrectal ultrasound. The safety profile of each procedure, which was determined by recording the incidence and nature of intraoperative and postoperative complications

Ethics statement:

The research protocol has been approved and reviewed by the Research Ethics Committee of the Faculty of Medicine, Ain Shams University. Written informed consent has been attained from all participants prior to enrolment, following a detailed explanation of the research's objectives, potential risks, procedures, and benefits. Participant confidentiality and data privacy were strictly maintained throughout all phases of the study. Participation was entirely voluntary, and individuals were informed of their right to withdraw from the study at any time without any consequences to their medical care

Statistical Analysis:

Statistical analysis was performed using IBM SPSS (Statistical Package for the social sciences) Statistics for Windows, Version 27.0 (IBM Corp., Armonk, USA). Continuous variables were expressed as mean ± standard deviation, and categorical variables as frequencies and percentages. Between-group comparisons were conducted using the Student's t-test for normally distributed continuous variables. The Chi-square (χ²) test or Fisher's exact test was applied for categorical variables, depending on expected cell counts. A two-tailed p-value < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lower urinary tract symptoms (voiding ± storage) refractory to medical treatment with IPSS > 20 (International Prostate Symptom Score) and Qmax < 15 mL/sec
* Refractory acute urinary retention
* Hematuria or recurrent urinary tract infections secondary to BPH
* Renal impairment secondary to prostatic obstruction

Exclusion Criteria:

* Proven malignancy by biopsy
* Urethral strictures
* Urinary bladder stones
* Previous prostate surgery
* Urodynamically proven neurogenic bladder
* Bladder cancer
* Unfit for anesthesia

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male participants only (self-identified
Enrollment: 56 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Maximum urinary flow rate (Qmax) at 12 months | Baseline and 12 months
  Mean change in maximum urinary flow rate (mL/sec) measured by uroflowmetry compared to baseline.

SECONDARY OUTCOMES:
Change in International Prostate Symptom Score (IPSS) from baseline to 12 months | 1 year
  Mean change in patient-reported IPSS questionnaire score compared to baseline, reflecting severity of lower urinary tract symptoms.
Operative time (minutes) | 1 year
  Duration of surgery measured in minutes from initial cystoscope insertion to removal.
Length of hospital stay (days) | Postoperative hospital stay
  Number of days from admission to discharge following surgery.
Duration of catheterization (days) | Postoperative period until catheter removal
  Total number of days patient remained catheterized postoperatively.
Post-void residual urine volume (PVR) at 12 months | Baseline and 12 months
  Mean post-void residual urine volume (mL) measured by ultrasound compared to baseline.
Serum prostate-specific antigen (PSA) at 12 months | Baseline and 12 months
  Mean change in serum PSA level (ng/mL) compared to baseline.
Residual prostate volume by transrectal ultrasound (TRUS) at 12 months | Baseline and 12 months
  Mean residual prostate volume (mL) measured by TRUS compared to baseline.
Number of participants with intraoperative and postoperative complications | ntraoperative and up to 12 months postoperative
  Frequency and type of complications recorded up to 12 months postoperatively, classified according to Clavien-Dindo system.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university _faculty of medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: https://sperlingprostatecenter.com/focal-laser-treatment-benign-prostatic-hyperplasia-bph/> — https://sperlingprostatecenter.com/focal-laser